CLINICAL TRIAL: NCT07096154
Title: Improving Emotional Wellbeing of University Students Using Culturally Adapted Cognitive Behavioural Approaches in Group Settings" (UniWELL-C): Protocol of a Feasibility and Effectiveness Study
Brief Title: Improving Emotional Wellbeing of University Students: Anxiety Management
Acronym: UniWELL-C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bogazici University (Other)
Responsible Party: Principal Investigator, Ayse Akan, Assistant Professor and Clinical Psychologist, Bogazici University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAP20022SUP
Record Dates: First submitted 2025-04-14; First posted 2025-07-31 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Anxiety
Keywords: anxiety; group therapy; CBT; university student mental health; mental health; cultural adapted psychotherapy
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Single-centre interventional non-blinded mixed-methods non-randomised pre-post design with a waitlist control and 6 weeks follow-up feasibility and psychotherapy effectiveness study.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT Experimental Arm (Experimental): An 8-session Group Cognitive Behavioural Therapy for anxiety management will be offered to the experimental group of about 40 university students who volunteered and scored above the threshold on the Beck Anxiety Inventory.
  Interventions: Behavioral: Group CBT Anxiety Management
- CBT Waitlist Arm (No Intervention): CBT waitlist control

INTERVENTIONS:
Behavioral: Group CBT Anxiety Management — An 8-session Group Cognitive Behavioural Therapy for anxiety management.
  Other Names: CBT; Group CBT
  Arms: CBT Experimental Arm

SUMMARY:
University students' psychological well-being is a growing public health concern. The university period is a key time for psychological, social, and academic development, which can increase vulnerability to mental health difficulties. Research suggests that group-based Cognitive Behavioural Therapy (CBT) is an effective, cost-efficient option for promoting student well-being. However, tailored interventions that reflect the cultural and contextual needs of specific populations are more likely to be effective. Western-based models of therapy may not always align with the cultural norms and experiences of students in countries like Türkiye.

In Türkiye, publicly accessible mental health services are limited, often reduced to short psychiatric consultations. Psychological therapies are primarily accessed privately, making free or low-cost university mental health services particularly valuable. Therefore, culturally adapted group CBT interventions may play a crucial role in supporting student mental health. This study, part of a larger project, aims to evaluate the effectiveness of CBT-based anxiety groups specifically tailored for Turkish university students.

Eligible participants are Bogazici University students aged 18 and over. Exclusion criteria include severe mental illness, high risk of harm to self or others, or scoring below the threshold on the Beck Anxiety Inventory. These individuals may require more specialized, individual support. The study includes participation in an 8-session CBT-based group focused on anxiety management. Participants may benefit from free psychological support, peer connection, and professional guidance. The study also contributes to the scientific literature by assessing the effectiveness of culturally adapted group interventions.

There are risks: participants may experience distress during sessions or while completing questionnaires. Support will be available from a master's student and/or the group therapist, under the supervision of a qualified clinical psychologist. If a participant's risk increases, they will be supported in accessing psychiatric care. An emergency contact will be required for safety. The study will run at Bogazici University in collaboration with BUREM and the Translational Clinical Psychology Lab, led by Dr. Ayse Akan (t-clinpsylab@bogazici.edu.tr). It is partially funded by Bogazici Scientific Research Projects (20022) and is expected to run for 1-3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a Bogazici University student.
2. Must be 18 years or older.
3. Must score above the threshold on the Beck Anxiety Inventory.

Exclusion Criteria:

1. Not Bogazici University student.
2. Has serious and severe mental illness.
3. High risk of self-harm/harm to others.
4. Scoring below the threshold of the Beck Anxiety Inventory.
5. Younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-07-03 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Beck Anxiety Inventory (BAI) | Baseline, immediately after the intervention, and follow-up 6 weeks after the completion of the intervention
  The Beck Anxiety Inventory (BAI) is a self-report questionnaire that measures the severity of anxiety levels. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severely - it bothered me a lot) resulting in a total score ranging from 0 to 63. Higher scores indicate greater levels of anxiety. The severity is categorized into "minimal", "mild", "moderate", and "severe".

SECONDARY OUTCOMES:
Depression Anxiety and Stress Scale (DASS42) | Baseline, immediately after the intervention, and follow-up 6 weeks after the completion of the intervention
  Depression Anxiety Stress Scale (DASS-42) is a questionnaire that measures the negative emotional states depression, anxiety and stress. Each subscale is scored separately. Each item is rated on a 4-point Likert scale from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). Scores for each subscale range from 0 to 42, and the combined total scale ranges from 0 to 126. Higher scores indicate more severity. The severity is categorized into "normal", "mild", "moderate", "severe", and "extremely severe".
Generalised Anxiety Disorder-7 (GAD7) | Baseline, immediately after the intervention, and follow-up 6 weeks after the completion of the intervention
  The Generalised Anxiety Disorder - 7 Scale (GAD7) is a questionnaire used to screen for Generalised Anxiety Disorder and assess the severity of anxiety symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day), resulting in a total score ranging from 0 to 21. Higher scores indicate more severity. The severity is categorized into "minimal", "mild", "moderate", and "severe".
Patient Health Questionnaire (PHQ9) | Baseline, immediately after the intervention, and follow-up 6 weeks after the completion of the intervention
  The Patient Health Questionnaire (PHQ9) is a scale used for assessing the presence and the severity of depression. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day), resulting in a total score that ranges from 0 to 27. Higher scores indicate more severity of depressive symptoms. The severity is categorized into "minimal", "mild", "moderate", "moderately severe" and "severe".
Outcome Rating Scale (ORS) | From enrollment to the end of treatment at 8 weeks
  Outcome Rating Scale (ORS) is a brief 4-item scale used for assessing the members' overall functioning in key areas: individual well-being, interpersonal relationships, social role, and overall well-being. Each item is rated on a visual analog scale from 0 to 10, resulting in a total score between 0 and 40. Higher scores indicate better overall functioning and well-being.
Qualitative data | Up to 12 weeks following the completion of the intervention
  Participants who completed their groups will also be invited to attend a semi-structured interview for in-depth qualitative feedback when they finish the intervention. Below are the sample questions to be asked to the participants:
  1. Could you tell us a little about the process (your mental health difficulties) that led you to apply to this group?
  2. Were you satisfied with the group?
  3. Which parts of the group were useful to you?
  4. Which parts of the group need to change (what you didn't like)?
  5. How was your relationship with the therapist and assistants?
  6. How was your relationship with the other participants of the group?
  7. What was the most important thing you learned from the group?
  8. Are there any other things that stood out to you?
  9. Would you recommend this group to other students with similar problems?
  10. Do you think this group should be an ongoing service provided by the university?

OTHER OUTCOMES:
Group Session Rating Scale (GSRS) | From enrollment to the end of treatment at 8 weeks
  Group Session Rating Scale (GSRS) is a brief 4-item scale used for assessing the members' evaluation of each session regarding the therapeutic relationship, goals and topics, approach or method, and overall experience. Each item is rated on a visual analog scale from 0 to 10, resulting in a total score between 0 and 40. Higher scores indicate more satisfaction with the group session.
Feedback Form | Immediately after the intervention
  The client feedback form is a 4-point self-report scale with a free-text box for additional comments. It is used to gather information about participants' experiences with the group facilitator and the intervention. The form includes questions about the therapeutic process, the structure of the sessions, the therapist's approach, and whether the support was helpful.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Akan, DClinPsych, Principal Investigator — Bogazici University
Locations (2):
- Turkey (Türkiye) (2):
  - Bogazici University Student Guidance and Psychological Counselling Centre (BUREM), Istanbul
  - Translational Clinical Psychology Lab, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
The anonymised quantitative data will be kept securely on a password protected drive for 10 years and will be shared with peer-reviewers if requested, while the qualitative interview transcripts will also be kept securely on a password protected drive but they will not be shared with peer-reviewers (will be only open to the research team) until it is deleted after 10 years. Some of the research team may use these data in secondary analysis projects.
Time Frame: The data supporting this study's findings will be available from the corresponding author upon reasonable request, starting immediately after publication. Data will be maintained and available for 10 years after the last data collection.
Access Criteria: Being a peer-reviewer / researcher